CLINICAL TRIAL: NCT01438060
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Flexible Dose Study of Aripiprazole in the Treatment of Patients With Psychosis Associated With Dementia of Alzheimer's Type
Brief Title: Aripiprazole in the Treatment of Patients With Psychosis Associated With Dementia of Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN138-006
Record Dates: First submitted 2011-09-02; First posted 2011-09-21 (Estimated); Results first posted 2012-03-05 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Dementia, Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole (BMS-337039) (Experimental): Double blind Acute Phase (Week 1 to Week 10), Open label Extension Phase (Week 11 to Week 140)
  Interventions: Drug: Aripiprazole (BMS-337039)
- Placebo (Placebo Comparator): Double blind Acute Phase (Week 1 to Week 10)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole (BMS-337039) — Acute Phase: Oral, Tablets (1 and 5 mg), Week 1-2: 2 mg, Week 3-4: 2 - 5 mg, Week 5-6: 2 - 10 mg, Weeks 7-10: 2 - 15 mg, Once daily, 10 weeks
  Extension Phase: Oral, Tablets (1 and 5 mg), Week 11: 2 mg, Weeks 12-13: 2 - 5 mg, Weeks 14-15: 2 - 10 mg, Weeks 16-140: 2 - 15 mg, Once daily, 130 weeks
  Arms: Aripiprazole (BMS-337039)
Drug: Placebo — Acute Phase: Oral, Tablets, 0 mg, Once daily, 10 Weeks
  Arms: Placebo

SUMMARY:
The primary objective of the study is to compare the efficacy of aripiprazole with placebo in patients with psychosis associated with Alzheimer's dementia.

DETAILED DESCRIPTION:
Open label Extension Phase: The 130-week Extension Phase was conducted to provide information regarding long-term safety and efficacy of aripiprazole in participants who were diagnosed at the onset of the Acute Phase with psychotic symptoms associated with dementia of the Alzheimer's type who responded to treatment in the 10-week Acute Phase of this study.

Treatment beyond 140 week: A country-specific amendment for France, allowed participants treated with aripiprazole who, according to the investigator's opinion, showed improvement at the Week 140 visit to continue treatment beyond 140 weeks. The termination was to be determined by clinical benefit to he participant.

Study design:

Acute Phase: Randomized, double-blind, placebo-controlled, flexible-dose, parallel-group study.

Extension Phase: Open label; flexible-dose.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized patients with a diagnosis of Alzheimer's disease as defined by Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV) criteria with symptoms of delusions or hallucinations, which have been present, at least intermittently for one month or longer
* Mini Mental State Examination (MMSE) score of 6 to 24 points
* Patients capable of self locomotion or locomotion with the aid of an assistive device
* Patients with an identified caregiver or proxy

For Extension Phase:

Eligible patients were males and females who had completed the 10-week Acute Phase in either treatment group; had a Week 10 Total Score of ≥ 6 on the NPI; and were, in the judgment of the investigator, deemed suitable for participation in the long-term trial.

Treatment beyond 140 weeks:

All subjects who completed the extension phase of CN138-006 in any French Investigational Site may be considered eligible for entry until they are no longer receiving clinical benefit, per the investigator's judgment

Exclusion Criteria:

* Patients with an Axis I (DSM IV) diagnosis of:

  * delirium
  * amnestic disorders
  * bipolar disorder
  * schizophrenia or schizoaffective disorder
  * mood disorder with psychotic features
* Patients with reversible causes of dementia
* Patients with psychotic symptoms continuously present since prior to the onset of the symptoms of dementia
* Patients with psychotic symptoms that are better accounted for by another general medical condition or by direct physiological effects of a substance
* Patients with a current major depressive episode with psychotic symptoms of hallucinations or delusions
* Patients with a diagnosis of dementia related to infection with the human immunodeficiency virus
* Patients with substance-induced persistent dementia
* Patients with dementia due to vascular causes, multi-infarct, head trauma, Pick's disease, Parkinson's disease, frontal or temporal dementia, Lewy body dementia, or any specific non-Alzheimer's type dementia
* Patients with seizure disorders
* Patients who have been refractory to neuroleptics used to treat psychotic symptoms in the past when treated for an adequate period with a therapeutic dose, unless permission is obtained from Bristol-Myers Squibb
* Patients who have met DSM-IV criteria for any significant substance use disorder within the 6 months prior to the start of screening

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2000-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 232 participants were enrolled, 24 were not randomized (baseline failures).
Groups:
- Placebo: Acute Phase: 0 mg, Once daily (10 Weeks)
- Aripiprazole: Acute Phase: Dosed at 2 mg/day (Week 1-2), 2-5 mg/day (Week 3-4), 2-10 mg/day (Week 5-6), 2-15 mg/day (Weeks 7-10).
Period: Acute Phase: Double-blind, 10 Weeks
Arm/Group | Placebo | Aripiprazole
Started | 102 | 106
Completed | 84 | 88
Not Completed | 18 | 18
Not completed — Adverse Event | 7 | 9
Not completed — Lack of Efficacy | 6 | 3
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 2
Not completed — Other Reason | 1 | 0
Period: Extension Phase: Week 10 to Week 130
Arm/Group | Placebo | Aripiprazole
Started | 80 (80 out of the 84 participants entered extension phase. All were treated with open-label aripiprazole) | 81 (Of the 88 participants, who completed Acute Phase, 81 opted to enter 130-week extension phase)
Completed | 22 | 25
Not Completed | 58 | 56
Not completed — Adverse Event | 15 | 16
Not completed — Lack of Efficacy | 8 | 8
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Participant Unreliability | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 22 | 12
Not completed — Other Reason | 7 | 15
Period: On Study Beyond Week 140
Arm/Group | Placebo | Aripiprazole
Started | 0 | 9 (9 participants in France who showed improvement at Week 140 continued treatment beyond 140 weeks)
Completed | 0 | 1
Not Completed | 0 | 8
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1
Not completed — Other Reason | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aripiprazole | Total
Number analyzed (Participants) | 102 | 106 | 208
Age Continuous [Median (Full Range); unit: years] | 82.0 [59 to 99] | 81.0 [56 to 95] | 81.0 [56 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 149
  Male | 28 | 31 | 59
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 98 | 105 | 203
  Black | 2 | 1 | 3
  Asian/ Pacific Islander | 2 | 0 | 2
Weight [Median (Full Range); unit: kg] | 58.8 [33 to 102] | 59.0 [35 to 100] | 59.0 [33 to 102]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Psychosis Subscale Score at Week 10 in Acute Phase
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 behavioral domains there are 4 scores: Frequency (scale:1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing).The NPI Psychosis Subscale consists of the two domains of Delusions and Hallucinations, calculated by adding the Individual Item Scores, to yield a possible total score of 0 to 24. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline (Day 0), Week 10
Population: Last Observation Carried forward (LOCF) data set, efficacy sample.
  Of the 208 randomized participants, 5 were excluded from the efficacy data sample: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2)
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Placebo: Acute Phase: 0 mg, Once daily (10 Weeks
- Aripiprazole: Acute Phase: 2 mg/day (Week 1-2), 2-5 mg/day (Week 3-4), 2-10 mg/day (Week 5-6), 2-15 mg/day (Weeks 7-10).
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a scale
  Baseline (Day 0) | 12.12 (0.60) | 12.29 (0.59)
  Mean Change from Baseline at Week 10 | -5.52 (0.66) | -6.55 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Analysis at Baseline (Day 0); Test type: Superiority or Other; p = 0.802, ANOVA — Baseline data was evaluated by analysis of variance (ANOVA) with treatment and study center as main effects; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-1.15 to 1.49] — Model based estimate
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Analysis at Week 10; Test type: Superiority or Other; p = 0.169, ANCOVA — ANCOVA model for LOCF data set included the baseline measure as covariate and the study center and treatment as main effects; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-2.49 to 0.44] — Model based estimate

2. Secondary Outcome: Change From Baseline in NPI Psychosis Subscale Score Through Week 8 in Acute Phase
Description: as for outcome 1
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, and 8
Population: LOCF data set, efficacy sample.
  Of the 208 randomized participants, 5 were excluded from the efficacy data sample: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2)
Measure: Mean (95% Confidence Interval); unit: Units on Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on Scale
  Baseline (Day 0) | 12.12 (0.60) [10.95 to 13.30] | 12.29 (0.59) [11.12 to 13.46]
  Week 1 | -3.33 (0.53) [-4.37 to -2.28] | -2.26 (0.52) [-3.29 to -1.22]
  Week 2 | -3.96 (0.67) [-5.27 to -2.65] | -3.81 (0.66) [-5.11 to -2.50]
  Week 3 | -4.54 (0.64) [-5.80 to -3.28] | -4.86 (0.64) [-6.12 to -3.61]
  Week 4 | -5.38 (0.61) [-6.59 to -4.18] | -5.66 (0.61) [-6.86 to -4.47]
  Week 6 | -4.87 (0.64) [-6.13 to -3.61] | -6.00 (0.63) [-7.25 to -4.75]
  Week 8 | -5.04 (0.69) [-6.40 to -3.69] | -6.01 (0.68) [-7.36 to -4.67]

3. Secondary Outcome: Change From Baseline in NPI Total Score in Acute Phase
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 behavioral domains there are 4 scores: Frequency (scale: 1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing).The NPI Total Score is calculated by adding the Individual Item Scores for all 12 domains, to yield a possible NPI Total Score of 0 to 144. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 40.08 (1.88) [36.38 to 43.78] | 39.82 (1.86) [36.14 to 43.49]
  Week 1 | -6.26 (1.58) [-9.39 to -3.13] | -4.13 (1.57) [-7.23 to -1.03]
  Week 2 | -9.98 (1.86) [-13.65 to -6.32] | -8.40 (1.84) [-12.04 to -4.77]
  Week 3 | -10.85 (2.13) [-15.04 to -6.65] | -8.61 (2.11) [-12.77 to -4.45]
  Week 4 | -11.81 (1.87) [-15.50 to -8.12] | -11.74 (1.86) [-15.40 to -8.08]
  Week 6 | -10.47 (2.09) [-14.59 to -6.35] | -11.61 (2.07) [-15.69 to -7.52]
  Week 8 | -9.68 (2.32) [-14.26 to -5.09] | -10.71 (2.30) [-15.26 to -6.17]
  Week 10 | -9.75 (2.35) [-14.40 to -5.11] | -11.20 (2.33) [-15.80 to -6.59]

4. Secondary Outcome: Participants Who Demonstrated a ≥ 50% Decrease From Baseline to Endpoint in the NPI Psychosis Subscale Score in Acute Phase
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Participants
  Week 1 | 24 | 18
  Week 2 | 37 | 34
  Week 3 | 45 | 44
  Week 4 | 52 | 47
  Week 6 | 53 | 56
  Week 8 | 58 | 64
  Week 10 | 60 | 70
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Analysis at Week 1; Test type: Superiority or Other; p = 0.391, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test with controlling for treatment and study center; Response ratio = 0.79, 95% CI 2-sided [0.47 to 1.35]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Analysis at Week 2; Test type: Superiority or Other; p = 0.766, Cochran-Mantel-Haenszel; CMH test with controlling for treatment and study center; Response ratio = 0.95, 95% CI 2-sided [0.69 to 1.31]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Analysis at Week 3; Test type: Superiority or Other; p = 0.967, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 1.01, 95% CI 2-sided [0.76 to 1.32]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Analysis at Week 4; Test type: Superiority or Other; p = 0.505, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 0.92, 95% CI 2-sided [0.71 to 1.19]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Analysis at Week 6; Test type: Superiority or Other; p = 0.590, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 1.07, 95% CI 2-sided [0.84 to 1.36]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Analysis at Week 8; Test type: Superiority or Other; p = 0.374, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 1.10, 95% CI 2-sided [0.89 to 1.37]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Analysis at Week 10; Test type: Superiority or Other; p = 0.175, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 1.15, 95% CI 2-sided [0.94 to 1.41]

5. Secondary Outcome: Participants Who Demonstrated a ≥ 50% Decrease From Baseline in the Total NPI Score in Acute Phase
Description: as for outcome 3
Time Frame: Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Participants
  Week 1 | 12 | 11
  Week 2 | 31 | 29
  Week 3 | 35 | 33
  Week 4 | 44 | 37
  Week 6 | 45 | 45
  Week 8 | 52 | 50
  Week 10 | 47 | 53
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Analysis at week 1; Test type: Superiority or Other; p = 0.753, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 0.88, 95% CI 2-sided [0.41 to 1.92]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Analysis at week 2; Test type: Superiority or Other; p = 0.600, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 0.90, 95% CI 2-sided [0.62 to 1.32]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Analysis at week 3; Test type: Superiority or Other; p = 0.673, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 0.93, 95% CI 2-sided [0.65 to 1.31]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Analysis at week 4; Test type: Superiority or Other; p = 0.255, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 0.83, 95% CI 2-sided [0.60 to 1.14]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Analysis at week 6; Test type: Superiority or Other; p = 0.958, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 0.99, 95% CI 2-sided [0.74 to 1.33]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Analysis at week 8; Test type: Superiority or Other; p = 0.525, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 0.92, 95% CI 2-sided [0.71 to 1.19]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Analysis at week 10; Test type: Superiority or Other; p = 0.602, Cochran-Mantel-Haenszel — CMH test with controlling for treatment and study center; Response ratio = 1.07, 95% CI 2-sided [0.82 to 1.40]

6. Secondary Outcome: Change From Baseline in NPI Psychosis Subscale Caregiver Distress Score in Acute Phase
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 behavioral domains there are 4 scores: Frequency (scale:1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale:0=not at all distressing to 5=extremely distressing). The NPI Psychosis Subscale Caregiver Distress Score is calculated by adding Individual Item Scores for the domains of Delusions and Hallucinations, to yield a possible total score of 0 to 10. Lower score=less severity. A negative change score from baseline=improvement.
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Unit on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Unit on a Scale
  Baseline (Day 0) | 4.80 (0.25) [4.30 to 5.29] | 4.70 (0.25) [4.21 to 5.19]
  Week 1 | -0.80 (0.21) [-1.21 to -0.38] | -0.64 (0.21) [-1.05 to -0.24]
  Week 2 | -0.84 (0.23) [-1.30 to -0.38] | -0.78 (0.23) [-1.24 to -0.33]
  Week 3 | -1.15 (0.24) [-1.62 to -0.69] | -0.93 (0.23) [-1.40 to -0.47]
  Week 4 | -1.31 (0.23) [-1.76 to -0.86] | -1.28 (0.23) [-1.73 to -0.84]
  Week 6 | -1.36 (0.27) [-1.89 to -0.84] | -1.62 (0.26) [-2.14 to -1.10]
  Week 8 | -1.18 (0.27) [-1.71 to -0.65] | -1.65 (0.27) [-2.17 to -1.12]
  Week 10 | -1.35 (0.26) [-1.86 to -0.83] | -1.79 (0.26) [-2.30 to -1.28]

7. Secondary Outcome: Change From Baseline in NPI Total Caregiver Distress Score in Acute Phase
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 behavioral domains there are 4 scores: Frequency (scale: 1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing).The total NPI Caregiver Distress Score is calculated by adding the 12 Caregiver Distress Individual Item Scores, to yield a possible total score of 0 to 60. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 16.58 (0.87) [14.87 to 18.29] | 17.06 (0.86) [15.37 to 18.76]
  Week 1 | -1.81 (0.65) [-3.08 to -0.53] | -1.64 (0.65) [-2.92 to -0.36]
  Week 2 | -3.25 (0.72) [-4.67 to -1.83] | -3.04 (0.72) [-4.47 to -1.61]
  Week 3 | -4.10 (0.81) [-5.76 to -2.44] | -2.58 (0.84) [-4.25 to -0.92]
  Week 4 | -4.01 (0.80) [-5.59 to -2.44] | -3.48 (0.80) [-5.06 to -1.90]
  Week 6 | -3.58 (0.98) [-5.51 to -1.66] | -3.72 (0.98) [-5.65 to -1.79]
  Week 8 | -3.20 (0.99) [-5.16 to -1.25] | -3.46 (0.99) [-5.42 to -1.50]
  Week 10 | -3.15 (1.03) [-5.19 to -1.11] | -3.53 (1.04) [-5.57 to -1.48]

8. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Severity of Illness Score in Acute Phase
Description: The CGI rating scale, which measures symptom severity, treatment response and the efficacy of treatments, is used in clinical studies on mental disorders. CGI Severity scale is a 7-point scale that requires the clinician to rate the severity of the illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. The assessment is based on severity of mental illness at the time of rating, 0=not assessed, 1=normal, 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill.
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: LOCF data set, efficacy sample.
  Of the 208 randomized participants, 5 were excluded from the efficacy data sample: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2). An additional participant did not have CGI-Severity score and was not included in the analysis
Measure: Mean (95% Confidence Interval); unit: Units on Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 102
Units on Scale
  Baseline (Day 0) | 4.84 (0.09) [4.67 to 5.01] | 4.83 (0.09) [4.66 to 5.00]
  Week 1 | -0.19 (0.08) [-0.34 to -0.04] | -0.10 (0.08) [-0.25 to 0.05]
  Week 2 | -0.29 (0.11) [-0.52 to -0.06] | -0.19 (0.12) [-0.41 to 0.04]
  Week 3 | -0.44 (0.11) [-0.65 to -0.22] | -0.44 (0.11) [-0.65 to -0.22]
  Week 4 | -0.47 (0.12) [-0.70 to -0.24] | -0.49 (0.12) [-0.73 to -0.26]
  Week 6 | -0.44 (0.12) [-0.69 to -0.20] | -0.58 (0.12) [-0.83 to -0.34]
  Week 8 | -0.56 (0.13) [-0.83 to -0.30] | -0.65 (0.13) [-0.92 to -0.39]
  Week 10 | -0.54 (0.14) [-0.82 to -0.26] | -0.69 (0.14) [-0.98 to -0.41]

9. Secondary Outcome: CGI Improvement Score in Acute Phase
Description: The CGI rating scale, which measures symptom severity, treatment response and the efficacy of treatments, is used in clinical studies on mental disorders. CGI Improvement scale is a 7 point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Weeks 1, 2, 3, 4, 6, 8, and 10
Population: LOCF data set, efficacy sample. n = Participants who had both post baseline and baseline values.
  Of the 208 randomized participants, 5 were excluded from the efficacy data sample: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2)
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on Scale
  Week 1; n=98, 102 | 3.81 (0.09) [lower limit 0.09] | 3.96 (0.08)
  Week 2; n=98, 102 | 3.55 (0.11) | 3.71 (0.10)
  Week 3; n=100, 103 | 3.37 (0.12) | 3.49 (0.11)
  Week 4; n=100, 103 | 3.28 (0.12) | 3.32 (0.12)
  Week 6; n=100, 103 | 3.26 (0.12) | 3.23 (0.13)
  Week 8; n=100, 103 | 3.11 (0.14) | 3.16 (0.13)
  Week 10; n=100, 103 | 3.07 (0.15) | 3.17 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Analysis at Week 1; Test type: Superiority or Other; p = 0.133, Cochran-Mantel-Haenszel — CMH Row Means test with controlling for study center
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Analysis at Week 2; Test type: Superiority or Other; p = 0.282, Cochran-Mantel-Haenszel — CMH Row Means test with controlling for study center
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Analysis at Week 3; Test type: Superiority or Other; p = 0.571, Cochran-Mantel-Haenszel — CMH Row Means test with controlling for study center
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Analysis at Week 4; Test type: Superiority or Other; p = 0.895, Cochran-Mantel-Haenszel — CMH Row Means test with controlling for study center
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Analysis at Week 6; Test type: Superiority or Other; p = 0.817, Cochran-Mantel-Haenszel — CMH Row Means test with controlling for study center
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Analysis at Week 8; Test type: Superiority or Other; p = 0.795, Cochran-Mantel-Haenszel — CMH Row Means test with controlling for study center
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Analysis at Week 10; Test type: Superiority or Other; p = 0.564, Cochran-Mantel-Haenszel — CMH Row Means test with controlling for study center

10. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale (BPRS) Total Score in Acute Phase
Description: The BPRS is designed to measure clinical change in participants and is used as a global measure of psychopathology. The BPRS includes 18 items with items devoted to hallucinatory behavior, suspiciousness, unusual thought content, etc. BPRS is an 18-item clinician rated scale with 11 general symptom items, 5 positive-symptom items, and 2 negative symptom items scored on a 7-point scale (1=not present and 7=extremely severe), with higher score indicating greater severity of symptom. Total possible score range=18 to 126.
  A negative change score signifies improvement.
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: Unit on Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Unit on Scale
  Baseline (Day 0); n=95, 100 | 43.42 (1.32) [40.32 to 46.02] | 43.63 (1.28) [41.10 to 46.16]
  Week 2; n=87, 95 | -4.65 (0.95) [-6.54 to -2.77] | -5.82 (0.94) [-7.68 to -3.96]
  Week 4; n=95, 100 | -5.80 (0.97) [-7.72 to -3.88] | -7.44 (0.95) [-9.31 to -5.58]
  Week 6; n=95, 100 | -6.13 (1.09) [-8.29 to -3.97] | -8.50 (1.07) [-10.60 to -6.40]
  Week 8; n=95, 100 | -6.45 (1.17) [-8.76 to -4.14] | -8.47 (1.14) [-10.72 to -6.22]
  Week 10; n=95, 100 | -6.28 (1.26) [-9.07 to -4.09] | -8.53 (1.23) [-10.95 to -6.10]

11. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score in Acute Phase
Description: The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language). It is a 19 item scale, the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
Time Frame: Baseline (Day 0), Week 10
Population: LOCF data set, efficacy sample. n=Participants who had both post baseline and baseline values.
  Of the 208 randomized participants, 5 were excluded from the efficacy data set: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2)
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on Scale
  Baseline (Day 0); N=86,94 | 14.13 (0.60) | 14.35 (0.58)
  Week 10; n=82, 87 | 0.53 (0.37) | -0.81 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Analysis at baseline; Test type: Superiority or Other; p = 0.733, ANCOVA; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-1.08 to 1.54]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Analysis at Week 10; Test type: Superiority or Other; p = 0.001, ANOVA; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-2.16 to -0.54]

12. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Delusions
Description: The 12 individual items in NPI that quantify behavioral changes in dementia are delusions, hallucinations, agitation, depression, anxiety, apathy, disinhibition, irritability, euphoria, aberrant motor behavior, nighttime behaviors, and appetite. For each behavioral domain there are 4 scores (refer to outcome 1 for the scoring for frequency, severity, total, caregiver distress). Presence of symptoms (0=no, 1=yes) x ratings for frequency and severity yield a total possible score of 0 to 12 for each item. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 7.85 [7.29 to 8.41] | 8.11 [7.55 to 8.67]
  Week 1 | -2.37 [-3.02 to -1.71] | -1.61 [-2.25 to -0.97]
  Week 2 | -2.84 [-3.69 to -1.98] | -2.72 [-3.57 to -1.88]
  Week 3 | -3.25 [-4.07 to -2.42] | -3.50 [-4.32 to -2.69]
  Week 4 | -3.72 [-4.54 to -2.90] | -3.89 [-4.69 to -3.08]
  Week 6 | -3.45 [-4.28 to -2.61] | -3.95 [-4.78 to -3.13]
  Week 8 | -3.52 [-4.41 to -2.63] | -3.91 [-4.79 to -3.03]
  Week 10 | -3.94 [-4.81 to -3.07] | -4.28 [-5.14 to -3.43]

13. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Hallucinations
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 4.27 [3.25 to 5.29] | 4.18 [3.17 to 5.19]
  Week 1 | -0.98 [-1.63 to -0.32] | -0.65 [-1.30 to 0.00]
  Week 2 | -1.15 [-1.86 to -0.43] | -1.09 [-1.80 to -0.38]
  Week 3 | -1.34 [-2.05 to -0.63] | -1.37 [-2.08 to -0.67]
  Week 4 | -1.71 [-2.31 to -1.10] | -1.79 [-2.40 to -1.19]
  Week 6 | -1.43 [-2.02 to -0.84] | -2.03 [-2.62 to -1.45]
  Week 8 | -1.57 [-2.22 to -0.91] | -2.12 [-2.77 to -1.47]
  Week 10 | -1.65 [-2.28 to -1.03] | -2.30 [-2.92 to -1.67]

14. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Agitation/Aggression
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 3.52 [2.68 to 4.37] | 4.04 [3.20 to 4.87]
  Week 1 | -0.34 [-1.12 to 0.43] | 0.10 [-0.68 to 0.88]
  Week 2 | -1.16 [-1.86 to -0.47] | -0.69 [-1.38 to 0.01]
  Week 3 | -0.73 [-1.50 to 0.03] | -0.59 [-1.35 to 0.17]
  Week 4 | -0.78 [-1.51 to -0.05] | -1.38 [-2.11 to -0.65]
  Week 6 | -0.31 [-1.08 to 0.46] | -0.94 [-1.71 to -0.18]
  Week 8 | -0.12 [-0.94 to 0.69] | -0.84 [-1.65 to -0.03]
  Week 10 | -0.47 [-1.32 to 0.37] | -1.12 [-1.96 to -0.28]

15. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Depression/Dysphoria
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 3.27 [2.59 to 3.95] | 2.28 [1.60 to 2.95]
  Week 1 | 0.21 [-0.39 to 0.81] | -0.04 [-0.62 to 0.54]
  Week 2 | -0.44 [-1.01 to 0.13] | -0.36 [-0.91 to 0.19]
  Week 3 | -0.77 [-1.28 to -0.25] | -0.33 [-0.84 to 0.17]
  Week 4 | -0.72 [-1.22 to -0.22] | -0.50 [-0.99 to -0.02]
  Week 6 | -0.47 [-1.04 to 0.10] | -0.55 [-1.10 to 0.00]
  Week 8 | -0.65 [-1.20 to -0.11] | -0.54 [-1.07 to -0.01]
  Week 10 | -0.32 [-0.95 to 0.32] | -0.42 [-1.04 to 0.19]

16. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Anxiety
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 3.64 [2.81 to 4.46] | 3.17 [2.36 to 3.99]
  Week 1 | 0.02 [-0.73 to 0.77] | 0.05 [-0.69 to 0.79]
  Week 2 | -0.08 [-0.73 to 0.58] | 0.08 [-0.56 to 0.72]
  Week 3 | -0.43 [-1.14 to 0.29] | 0.07 [-0.63 to 0.77]
  Week 4 | -0.80 [-1.47 to -0.14] | -0.38 [-1.03 to 0.27]
  Week 6 | -0.79 [-1.49 to -0.08] | -0.13 [-0.82 to 0.57]
  Week 8 | -0.23 [-0.90 to 0.44] | -0.21 [-0.87 to 0.46]
  Week 10 | -0.43 [-1.13 to 0.26] | -0.31 [-0.99 to 0.37]

17. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Apathy/Indifference
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 4.14 [3.41 to 4.86] | 3.47 [2.75 to 4.19]
  Week 1 | 0.03 [-0.66 to 0.71] | -0.70 [-1.37 to -0.03]
  Week 2 | -0.48 [-1.11 to 0.15] | -0.76 [-1.37 to -0.14]
  Week 3 | -0.09 [-0.80 to 0.62] | -0.36 [-1.06 to 0.33]
  Week 4 | -0.65 [-1.39 to 0.10] | -0.67 [-1.40 to 0.06]
  Week 6 | -0.63 [-1.43 to 0.17] | -0.40 [-1.18 to 0.38]
  Week 8 | -0.87 [-1.60 to -0.15] | -0.21 [-0.92 to 0.49]
  Week 10 | -0.95 [-1.78 to -0.11] | -0.09 [-0.91 to 0.72]

18. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Elation/Euphoria
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 0.56 [0.06 to 1.05] | 0.73 [0.24 to 1.23]
  Week 1 | -0.48 [-0.75 to -0.22] | -0.26 [-0.52 to 0.01]
  Week 2 | -0.37 [-0.63 to -0.11] | -0.18 [-0.43 to 0.08]
  Week 3 | -0.48 [-0.76 to -0.20] | -0.27 [-0.54 to 0.01]
  Week 4 | -0.47 [-0.66 to -0.28] | -0.40 [-0.59 to -0.21]
  Week 6 | -0.38 [-0.58 to -0.18] | -0.39 [-0.59 to -0.20]
  Week 8 | -0.32 [-0.59 to -0.04] | -0.25 [-0.52 to 0.03]
  Week 10 | -0.42 [-0.65 to -0.19] | -0.36 [-0.59 to -0.14]

19. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Disinhibition
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 0.98 [0.39 to 1.57] | 1.36 [0.77 to 1.94]
  Week 1 | -0.14 [-0.54 to 0.25] | -0.39 [-0.79 to 0.00]
  Week 2 | -0.42 [-0.91 to 0.07] | -0.44 [-0.93 to 0.05]
  Week 3 | -0.27 [-0.86 to 0.32] | -0.21 [-0.80 to 0.38]
  Week 4 | -0.55 [-1.04 to -0.06] | -0.67 [-1.16 to -0.19]
  Week 6 | -0.19 [-0.64 to 0.26] | -0.72 [-1.17 to -0.28]
  Week 8 | -0.20 [-0.67 to 0.28] | -0.44 [-0.91 to 0.03]
  Week 10 | 0.07 [-0.47 to 0.60] | -0.35 [-0.88 to 0.18]

20. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Irritability/Lability
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 3.73 [2.80 to 4.66] | 4.36 [3.44 to 5.28]
  Week 1 | -0.73 [-1.48 to 0.02] | -0.09 [-0.84 to 0.66]
  Week 2 | -0.89 [-1.65 to -0.12] | -0.69 [-1.45 to 0.08]
  Week 3 | -1.11 [-1.89 to -0.32] | -1.09 [-1.87 to -0.30]
  Week 4 | -0.75 [-1.53 to 0.02] | -1.53 [-2.30 to -0.76]
  Week 6 | -0.42 [-1.19 to 0.36] | -1.29 [-2.06 to -0.51]
  Week 8 | -0.33 [-1.16 to 0.50] | -0.99 [-1.82 to -0.16]
  Week 10 | -0.24 [-1.02 to 0.53] | -1.26 [-2.03 to -0.48]

21. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Aberrant Motor Behavior
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 3.67 [2.69 to 4.66] | 3.61 [2.63 to 4.59]
  Week 1 | -0.66 [-1.26 to -0.06] | 0.18 [-0.42 to 0.77]
  Week 2 | -0.84 [-1.63 to -0.06] | -0.51 [-1.29 to 0.27]
  Week 3 | -1.68 [-2.45 to -0.09] | -0.66 [-1.43 to 0.12]
  Week 4 | -0.91 [-1.73 to -0.09] | -0.16 [-0.98 to 0.65]
  Week 6 | -0.89 [-1.64 to -0.13] | -0.61 [-1.36 to 0.14]
  Week 8 | -1.06 [-1.78 to -0.33] | -0.83 [-1.55 to -0.11]
  Week 10 | -1.02 [-1.83 to -0.22] | -0.89 [-1.69 to -0.09]

22. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Appetite/Eating Behaviors
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 1.78 [1.18 to 2.39] | 1.47 [0.87 to 2.07]
  Week 1 | -0.24 [-0.73 to 0.25] | -0.18 [-0.66 to 0.30]
  Week 2 | -0.36 [-0.84 to 0.12] | -0.21 [-0.68 to 0.26]
  Week 3 | -0.14 [-0.65 to 0.36] | 0.23 [-0.27 to 0.73]
  Week 4 | -0.44 [-0.96 to 0.07] | -0.04 [-0.55 to 0.47]
  Week 6 | -0.27 [-0.96 to 0.42] | 0.23 [-0.45 to 0.91]
  Week 8 | -0.11 [-0.72 to 0.49] | 0.45 [-0.15 to 1.05]
  Week 10 | -0.17 [-0.79 to 0.46] | 0.56 [-0.05 to 1.17]

23. Secondary Outcome: Change From Baseline in NPI Individual Item Scores in Acute Phase: Sleep
Description: as for outcome 12
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on a Scale
  Baseline (Day 0) | 2.67 [1.78 to 3.55] | 3.03 [2.15 to 3.91]
  Week 1 | -0.10 [-0.84 to 0.64] | -0.07 [-0.81 to 0.67]
  Week 2 | -0.20 [-0.95 to 0.55] | -0.07 [-0.82 to 0.67]
  Week 3 | -0.20 [-0.98 to 0.58] | 0.10 [-0.68 to 0.87]
  Week 4 | 0.02 [-0.65 to 0.70] | 0.15 [-0.53 to 0.82]
  Week 6 | -0.39 [-1.12 to 0.34] | -0.03 [-0.76 to 0.69]
  Week 8 | -0.06 [-0.80 to 0.68] | -0.06 [-0.79 to 0.68]
  Week 10 | 0.05 [-0.69 to 0.79] | -0.06 [-0.80 to 0.67]

24. Secondary Outcome: Change From Baseline in Simpson-Angus Scale (SAS) Total Score in Acute Phase
Description: The SAS is a 10-item instrument used to evaluate the presence and severity of parkinsonian symptomatology. It is the most commonly used rating scale for Parkinsonism in clinical trials over the past 25 years. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The total SAS Score has a possible range from 10 to 50.(lower score=less severe). Negative change scores indicate improvement.
Time Frame: Baseline (Day 0), Weeks 2, 4, and 10
Population: Observed cases data set, Efficacy Sample. n=Participants who had both post baseline and baseline values.
  Of the 208 randomized participants, 5 were excluded from the efficacy data set: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2)
Measure: Mean (95% Confidence Interval); unit: Units on scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on scale
  Baseline (Day 0); n=97, 100 | 14.41 (NA) [13.37 to 15.46] | 14.47 (NA) [13.45 to 15.50]
  Week 2; n=89, 94 | 0.02 [-0.49 to 0.52] | -0.35 [-0.84 to 0.14]
  Week 4; n=93, 96 | -0.15 [-0.76 to 0.45] | -0.06 [-0.65 to 0.54]
  Week 10; n=82, 85 | -0.44 [-1.19 to 0.31] | 0.33 [-0.40 to 1.07]

25. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score in Acute Phase
Description: The Abnormal Involuntary Movement Scale (AIMS) is a rating scale that was designed to measure involuntary movements (tardive dyskinesia). The AIMS test has a total of twelve items rating involuntary movements of various areas of the patient's body. These items are rated on a five-point scale of severity from 0-4. The scale is rated from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe).
  AIMS Total Score is from 0 to 28. A negative change score signifies improvement.
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, and 10
Population: Observed Cased data set, efficacy sample. n=Participants who had both post baseline and baseline values.
  Of the 208 randomized participants, 5 were excluded from the efficacy data set: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2)
Measure: Mean (95% Confidence Interval); unit: Units on scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Units on scale
  Baseline (Day 0); n=99, 101 | 0.87 [0.32 to 1.42] | 0.93 [0.39 to 1.48]
  Week 2; n=91, 95 | -0.10 [-0.25 to 0.04] | -0.17 [-0.32 to -0.03]
  Week 4; n=97, 97 | -0.05 [-0.30 to 0.19] | -0.08 [-0.33 to 0.17]
  Week 8; n=87, 87 | 0.07 [-0.30 to 0.44] | -0.14 [-0.51 to 0.23]
  Week 10; n=85, 87 | 0.05 [-0.33 to 0.43] | -0.17 [-0.55 to 0.20]

26. Secondary Outcome: Change From Baseline in Barnes Global Clinical Assessment of Akathisia in Acute Phase
Description: The Barnes Akathisia Rating Scale is a 4-item scale to assess presence and severity of drug-induced akathisia, including both objective items and subjective items, together with a global clinical assessment of akathisia. Global assessment is made on a scale of 0 to 5 with comprehensive definitions provided for each anchor point on scale: 0=absent; 1=questionable; 2=mild akathisia; 3=moderate akathisia; 4=marked akathisia; 5=severe akathisia. Score has a possible range from 0 (absent) to 5 (severe akathisia). Negative change scores indicate improvement in akathisia.
Time Frame: Baseline (Day 0), Weeks 1, 2, 3, 4, 6, 8, and 10
Population: Observed cases data set, efficacy sample. n=Participants with both post-baseline and baseline measures.
  Of the 208 randomized participants, 5 were excluded from the efficacy data sample: 2 from placebo (Withdrew Consent, Inadequate Caregiver Input.); 3 in aripiprazole group (Withdrew Consent-1, AE-2)
Measure: Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 100 | 103
Unit on scale
  Baseline (Day 0); n=100,101 | 0.20 [0.09 to 0.31] | 0.19 [0.07 to 0.30]
  Week 1; n=99, 101 | -0.06 [-0.12 to 0.00] | -0.06 [-0.12 to 0.00]
  Week 2; n=91, 95 | -0.02 [-0.07 to 0.03] | -0.05 [-0.11 to 0.00]
  Week 3; n=95, 99 | -0.03 [-0.08 to 0.02] | -0.06 [-0.11 to -0.01]
  Week 4; n=97, 98 | 0.00 (NA) [-0.07 to 0.07] | -0.08 [-0.15 to -0.02]
  Week 6; n=91, 92 | -0.07 [-0.14 to -0.01] | -0.02 [-0.09 to 0.04]
  Week 8; n=87, 87 | -0.05 [-0.11 to 0.01] | -0.03 [-0.09 to 0.03]
  Week 10; n=85, 87 | -0.05 [-0.11 to 0.00] | -0.05 [-0.11 to 0.01]

27. Secondary Outcome: Participants With Extrapyramidal Symptoms (EPS) Related Adverse Events in Acute Phase
Description: Extrapyramidal symptoms (EPS) are various movement disorders such as acute dystonic reactions, pseudoparkinsonism, or akathisia
Time Frame: Week 1 to week 10
Population: Of the 208 randomized participants, one (randomized to aripiprazole) was excluded from the Safety Sample as the participant withdrew consent prior to receiving study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 102 | 105
Participants
  Dyskinesia | 2 | 0
  Extrapyramidal syndrome | 1 | 2
  Hypertonia | 1 | 1
  Hypokinesia | 0 | 1
  Tremor | 0 | 2

28. Secondary Outcome: Participants Who Died, Experienced Serious Adverse Events (SAEs), Adverse Events (AEs) or Discontinuations Due to AEs in Acute Phase
Description: AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a cancer, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Week 1 to week 10
Population: as for outcome 27
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 102 | 105
Participants
  Any adverse event (AE) | 53 | 67
  Serious adverse event | 9 | 16
  Deaths | 0 | 4
  Discontinuations due to AE | 7 | 11

29. Secondary Outcome: Participants With Potentially Clinically Significant Laboratory Abnormalities in Acute Phase
Description: Criteria for identifying potentially clinically significant laboratory values were based on guidelines suggested by the FDA Division of Neuropharmacological Drug Products. Normal ranges are local lab data and vary according to the site. M=male, F=female. Criteria for hematocrit also includes a 3 point shift from baseline.
Time Frame: Week 1 to Week 10
Population: Of the 208 randomized participants, one (randomized to aripiprazole) was excluded from the Safety Sample as the participant withdrew consent prior to receiving study medication. n=Participants with values for laboratory findings
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 102 | 105
Participants
  Alanine aminotransferase ≥3 x ULN; n=98, 98 | 1 | 3
  Aspartate aminotransferase ≥3 x ULN; n=98, 98 | 1 | 1
  Alkaline phosphatase ≥3 x ULN; n=98, 98 | 1 | 0
  Creatine phosphokinase (total) ≥3 x ULN; n=98, 98 | 1 | 2
  Creatinine ≥ 2.0 mg/dL; n=98, 98 | 2 | 2
  Uric acid ≥8.5 mg/dL (F);≥10.5 mg/dL(M); n=98, 98 | 5 | 2
  Calcium ≥ 10.6 mg/dL; n=98, 98 | 1 | 2
  Calcium ≤ 8.4 mg/dL; n=98, 98 | 4 | 5
  Serum Chloride ≥ 113 mEq/L; n=98, 98 | 6 | 4
  Serum Chloride ≤ 93 mEq/L; n=98, 98 | 5 | 6
  Cholesterol Total > ULN; n=98, 98 | 47 | 36
  Cholesterol Total < LLN; n=98, 98 | 1 | 0
  Serum Glucose Fasting > ULN; n=36, 31 | 13 | 16
  Serum Potassium ≥ 5.6 mEq/L; n=98, 98 | 7 | 7
  Serum Potassium ≤ 3.4 mEq/L; n=98, 98 | 4 | 4
  Serum Sodium ≥ 148 mEq/L; n=98, 98 | 2 | 1
  Serum Sodium ≤ 132 mEq/L; n=98, 98 | 3 | 3
  Urea ≥ 10.1mmol/L; n=98, 97 | 19 | 14
  Platelet ≥ 700,000 mm3; n=97, 96 | 0 | 1
  Platelet ≤ 75,000 mm3; n=97, 96 | 1 | 0
  Eosinophils ≥ 10%; n=97, 96 | 1 | 1
  Hematocrit ≤ 37% (M)/≤ 32% (F); n=97, 96 | 7 | 6
  Hemoglobin ≤ 11.5 (M)/≤ 9.5 g/dL (F); n=97, 96 | 6 | 4
  Urine Glucose ≥ 2-unit increase; n=92, 93 | 2 | 0
  Urine Protein ≥ 2-unit increase; n=92, 93 | 2 | 1

30. Secondary Outcome: Participants With Potentially Clinically Significant (PCS) Vital Sign Abnormalities in Acute Phase
Description: Systolic BP: increase defined as ≥180 and a ≥20-mmHg increase from baseline (BL); decrease defined as ≤90 and a ≥20mmHg decrease from BL. Diastolic BP: increase defined as ≥105 and a ≥15mmHg decrease from BL, decrease defined as ≤50 and a ≥15mmHg decrease from BL. Heart rate: increase defined as ≥120 and ≥15bpm increase from BL, decrease defined as ≤50 and ≥15bpm decrease from BL; Weight: increase defined as ≥7% from BL, decrease defined as ≤7% decrease BL. Criteria for identifying PCS measurements are based on guidelines suggested by the FDA Division of Neuropharmacological Drug Products
Time Frame: Week 1 to week 10
Population: Of the 208 randomized participants, one (randomized to aripiprazole) was excluded from the Safety Sample as the participant withdrew consent prior to receiving study medication. n=Participants with values for vital signs
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 102 | 105
Participants
  Increased Systolic BP, standing; n=99, 100 | 5 | 5
  Decreased Systolic BP, standing; n=99, 100 | 1 | 1
  Increased Systolic BP, supine; n=101, 102 | 6 | 2
  Decreased Systolic BP, supine; n=101, 102 | 0 | 2
  Decreased Systolic BP, sitting; n=13, 20 | 0 | 1
  Increased Diastolic BP, standing; n=99, 100 | 2 | 2
  Decreased Diastolic BP, standing; n=99, 100 | 6 | 3
  Increased Diastolic BP, supine; n=101, 102 | 2 | 0
  Decreased Diastolic BP, supine; n=101, 102 | 4 | 3
  Decreased Diastolic BP, sitting; n=13, 20 | 2 | 0
  Increased Heart rate, standing; n=99, 100 | 1 | 0
  Decreased Heart rate, standing; n=99, 100 | 0 | 1
  Decreased Heart rate, supine; n=101, 102 | 1 | 3
  Increased Weight; n=89, 93 | 3 | 5
  Decreased Weight; n=89,93 | 5 | 5

31. Secondary Outcome: Participants With Potentially Clinically Significant Electrocardiogram Abnormalities in Acute Phase
Description: Bradycardia:Heart rate ≤50 bpm and ≥15 bpm decrease from baseline; Supraventricular premature beat: ≥2 per 10 seconds and any increase from baseline; 1st degree A-V Block: PR ≥0.20 seconds and increase of ≥0.05 second from baseline; Intraventricular conduction block:QRS ≥0.12 second and increase of ≥0.02 second from baseline; QTcB= ≥450 msec and ≥10% increase from baseline; QTcN =≥450 msec and ≥10% increase from baseline. All other events were not present at baseline but observed during the study. Inc=increase
Time Frame: Week 1 to Week 10
Population: Of the 208 randomized participants, one (randomized to aripiprazole) was excluded from the Safety Sample as the participant withdrew consent prior to receiving study medication. n=Participants who were evaluated for electrocardiogram
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 102 | 105
Participants
  Bradycardia; n=99, 102 | 3 | 1
  Sinus Bradycardia; n=99, 102 | 2 | 1
  Supraventricular premature beat; n=99, 102 | 10 | 7
  Ventricular premature beat; n=99, 102 | 7 | 12
  Supraventricular tachycardia; n=99, 102 | 1 | 0
  Atrial fibrillation; n=99, 102 | 3 | 1
  Atrial flutter; n=99, 102 | 0 | 1
  1st degree A-V Block; n=95, 97 | 2 | 0
  Left bundle branch block; n=99, 102 | 1 | 2
  Right bundle branch block; n=99, 102 | 2 | 1
  Other intraventricular conduction block; n=99, 102 | 0 | 2
  Subacute infarction; n=99, 102 | 1 | 0
  Old infarction; n=99, 102 | 2 | 2
  Myocardial ischemia; n=99, 102 | 3 | 4
  Symmetrical T-wave inversion; n=99, 102 | 2 | 1
  Inc QTcB (≥450 msec≥,10% from baseline); n=99, 102 | 5 | 5
  Inc QTcN (≥450 msec,≥10% from baseline); n=99, 102 | 1 | 2

32. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI) Psychosis Subscale Score From Baseline During Extension Phase
Description: as for outcome 1
Time Frame: Baseline (Day 0), Weeks 18,26,40,52,68,84,100,116,132,140
Population: Observed Cases data set, Efficacy Sample. n=participants with both post-baseline and baseline values
  Of the 161 participants (80 in placebo and 81 in aripiprazole group), 158 were included in the Extension Phase Efficacy Sample, (3 treated participants had no efficacy measurements).
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- Aripiprazole: Aripiprazole dosed at 2 mg (Week 11), 2-5 mg/day (Weeks 12-13), 2-10 mg/day (Weeks 14-15), 2-15 mg/day (Weeks 16-140).
Arm/Group | Aripiprazole
Number analyzed (Participants) | 158
Units on a Scale
  Baseline, Day 0 (n=154) | 12.312 (0.426)
  Week 18 (n=151) | -8.589 (0.548)
  Week 26 (n=139) | -8.993 (0.589)
  Week 40 (n=115) | -8.270 (0.677)
  Week 52 (n=98) | -8.582 (0.672)
  Week 68 (n=69) | -9.232 (0.824)
  Week 84 (n=62) | -10.18 (0.848)
  Week 100 (n=52) | -10.06 (1.031)
  Week 116 (n=47) | -10.19 (1.183)
  Week 132 (n=31) | -11.68 (1.554)
  Week 140 (n=25) | -13.12 (1.586)

33. Secondary Outcome: Clinical Global Impression (CGI) Improvement Score During Extension Phase
Description: as for outcome 9
Time Frame: Weeks 12, 14, 18, 22, 26, 30, 34, 40, 46, 52, 68, 84, 100, 116, 132, 140
Population: Observed Cases data set, Efficacy Sample. n=participants with both post-baseline and baseline values.
  Of the 161 participants, 158 were included in the Extension Phase Efficacy Sample, (3 treated participants had no efficacy measurements).
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 158
Units on Scale
  Week 12; n=158 | 2.873 (0.089)
  Week 14; n=151 | 2.709 (0.084)
  Week 18; n=152 | 2.625 (0.091)
  Week 22; n=145 | 2.552 (0.087)
  Week 26; n=140 | 2.707 (0.113)
  Week 30; n=129 | 2.636 (0.113)
  Week 34; n=121 | 2.554 (0.106)
  Week 40; n=114 | 2.482 (0.121)
  Week 46; n=103 | 2.592 (0.130)
  Week 52; n=100 | 2.580 (0.138)
  Week 68; n=70 | 2.514 (0.155)
  Week 84; n=62 | 2.306 (0.150)
  Week 100; n=53 | 2.660 (0.196)
  Week 116; n=47 | 2.787 (0.233)
  Week 132; n=36 | 3.028 (0.289)
  Week 140; n=26 | 2.385 (0.299)

34. Secondary Outcome: Change in Abnormal Involuntary Movement Scale (AIMS) Total Score During Extension Phase
Description: AIMS is a rating scale that was designed to measure involuntary movements (tardive dyskinesia). The AIMS test has a total of twelve items rating involuntary movements of various areas of the patient's body. These items are rated on a five-point scale of severity from 0-4. The scale is rated from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe).
  AIMS Total Score is from 0 to 28. A negative change score signifies improvement.
Time Frame: End of Acute Phase (Week 10), Weeks 14, 18, 22, 26, 30, 34, 40, 46, 52, 68, 84, 100, 116, 140
Population: Observed Cases data set, Efficacy Sample. n=participants with both post-baseline and baseline values.
  Of the 161 participants (80 in placebo and 81 in aripiprazole group), 158 were included in the Extension Phase Efficacy Sample, (3 treated participants had no efficacy measurements).
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 158
Units on Scale
  End of Acute Phase (Week 10); n=157 | 0.95 (0.20)
  Week 14; n=151 | 0.25 (0.12)
  Week 18; n=152 | 0.09 (0.11)
  Week 22; n=145 | 0.02 (0.13)
  Week 26; n=140 | -0.12 (0.13)
  Week 30; n=128 | -0.01 (0.10)
  Week 34; n=121 | -0.10 (0.15)
  Week 40; n=115 | -0.01 (0.16)
  Week 46; n=104 | -0.02 (0.15)
  Week 52; n=100 | -0.02 (0.20)
  Week 68; n=70 | -0.29 (0.17)
  Week 84; n=62 | -0.24 (0.17)
  Week 100; n=52 | -0.21 (0.15)
  Week 116; n=47 | -0.21 (0.20)
  Week 140; n=15 | 0.00 (0.20)
  Endpoint (LOCF data set); n=157 | -0.03 (0.15)

35. Secondary Outcome: Change in Simpson-Angus Scale (SAS) Total Score During Extension Phase
Description: The SAS is a 10-item instrument used to evaluate the presence and severity of parkinsonian symptomatology. It is the most commonly used rating scale for Parkinsonism in clinical trials over the past 25 years. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The total SAS Score has a possible range from 10 to 50 (lower score=less severe). Negative change scores indicate improvement.
Time Frame: End of Acute Phase (Week 10), Weeks 18,26, 40, 52
Population: as for outcome 33
Measure: Mean (Standard Error); unit: Units on Scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 158
Units on Scale
  End of Acute Phase (Week 10); n=153 | 14.34 (0.40)
  Week 18; n=148 | 0.62 (0.23)
  Week 26; n=132 | 1.24 (0.31)
  Week 40; n=107 | 1.25 (0.39)
  Week 52; n=95 | 1.14 (0.40)
  Endpoint (LOCF data set); n=153 | 2.01 (0.37)

36. Secondary Outcome: Change in Barnes Global Clinical Assessment of Akathisia Score During Extension Phase
Description: as for outcome 26
Time Frame: End of Acute Phase (Week 10), Weeks 18,26, 40, 52
Population: as for outcome 33
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole
Number analyzed (Participants) | 158
units on a scale
  End of Acute Phase (Week 10); n=155 | 0.14 (0.03)
  Week 18; n=151 | 0.04 (0.03)
  Week 26; n=139 | 0.03 (0.04)
  Week 40; n=114 | 0.04 (0.04)
  Week 52; n=99 | 0.06 (0.03)
  Endpoint (LOCF data set); n=155 | 0.06 (0.03)

37. Secondary Outcome: Participants With Extrapyramidal Symptoms (EPS) Related Adverse Events During Extension Phase
Description: as for outcome 27
Time Frame: Week 11 to Week 140
Population: All the 161 participants (80 in placebo and 81 in aripiprazole group)were included in the Extension Phase Safety Sample.
Measure: Number; unit: Participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 161
Participants
  Dyskinesia | 2
  Muscle Rigidity | 3
  Extrapyramidal Disorder | 14
  Hypokinesia | 8
  Tremor | 8
  Akinesia | 1
  Bradykinesia | 1
  Parkinsonian Gait | 1
  Muscle Twitching | 1

38. Secondary Outcome: Participants Who Died, Experienced Serious Adverse Events (SAEs), Adverse Events (AEs) or Discontinuations Due to AE During Extension Phase
Description: as for outcome 28
Time Frame: Week 11 to Week 140
Population: All the 161 participants (80 in placebo and 81 in aripiprazole group)were included in the Extension Phase Safety Sample.
Measure: Number; unit: Participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 161
Participants
  Death | 41
  SAE | 59
  AE | 148
  Discontinuation due to AE | 66

39. Secondary Outcome: Participants With a Potentially Clinically Significant Vital Sign Abnormality During Extension Phase
Description: Systolic BP: increase defined as ≥180 and a ≥20-mmHg increase from baseline (BL); decrease defined as ≤90 and a ≤20mmHg decrease from BL. Diastolic BP: increase defined as ≥105 and a ≥15mmHg decrease from BL, decrease defined as ≤50 and a ≤15mmHg decrease from BL. Heart rate: increase defined as ≥120 and ≥15bpm increase from bBL, decrease defined as ≤50 and ≤15bpm decrease from BL; Weight: increase defined as ≥7% from baseline, decrease defined as ≤7% decrease BL. Criteria for identifying PCS measurements based on guidelines suggested by the FDA Division of Neuropharmacological Drug Products
Time Frame: Week 11 to Week 140
Population: All the 161 participants (80 in placebo and 81 in aripiprazole group) were included in the Extension Phase Safety Sample.
Measure: Number; unit: Participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 161
Participants
  Increased Systolic BP, standing; n=159 | 6
  Decreased Systolic BP, standing; n=159 | 9
  Increased Systolic BP, supine; n=158 | 6
  Decreased Systolic BP, supine; n=158 | 7
  Decreased Systolic BP, sitting; n=45 | 1
  Increased Diastolic BP, standing; n=159 | 4
  Decreased Diastolic BP, standing; n=159 | 19
  Increased Diastolic BP, supine; n=158 | 1
  Decreased Diastolic BP, supine; n=158 | 25
  Decreased Diastolic BP, sitting; n=45 | 1
  Increased Heart rate, standing; n=159 | 2
  Decreased Heart rate, standing; n=159 | 3
  Increased Heart rate, supine; n=158 | 1
  Decreased Heart rate, supine; n=158 | 5
  Increased Weight; n=133 | 28
  Decreased Weight; n=133 | 58

40. Secondary Outcome: Participants With a Potentially Clinically Significant Electrocardiogram Abnormalities During Extension Phase
Description: Bradycardia:Heart rate ≤50 bpm and ≥15 bpm decrease from baseline; Supraventricular premature beat: ≥2 per 10 seconds and any increase from baseline; 1st degree A-V Block: PR ≥0.20 seconds and increase of ≥0.05 second from baseline; Intraventricular conduction block:QRS ≥0.12 second and increase of ≥0.02 second from baseline; QTcB= ≥450 msec and ≥10% increase from baseline; QTcN =≥450 msec and ≥10% increase from baseline. All other events were not present at baseline but observed during the study
Time Frame: Week 11 to Week 140
Population: as for outcome 39
Measure: Number; unit: Participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 161
Participants
  Atrial Fibrillation; n=145 | 5
  Atrial Flutter; n=145 | 1
  Bradycardia; n=145 | 4
  Left Bundle Branch Block; n=145 | 5
  Myocardial Ischemia; n=145 | 10
  Old Infarction; n=145 | 2
  Right Bundle Branch Block; n=145 | 3
  Sinus Bradycardia; n=145 | 2
  Sinus Tachycardia; n=145 | 2
  Supraventricular Premature Beat; n=145 | 12
  Supraventricular Tachycardia; n=145 | 2
  Symmetrical T-wave Inversions; n=145 | 8
  Tachycardia; n=145 | 4
  Ventricular premature Beat; n=145 | 13

41. Secondary Outcome: Participants With Potentially Clinically Significant Laboratory Abnormalities During Extension Phase
Description: Criteria for identifying potentially clinically significant laboratory values were based on guidelines suggested by the FDA Division of Neuropharmacological Drug Products.
Time Frame: Week 11 to Week 140
Population: as for outcome 39
Measure: Number; unit: Participants
Arm/Group | Aripiprazole
Number analyzed (Participants) | 161
Participants
  High Alanine aminotransferase; ≥ 41 U/L | 0
  High Aspartate aminotransferase; ≥ 38 U/L | 1
  High Alkaline phosphatase; ≥ 117 U/L | 2
  High Lactate dehydrogenase; >480 U/L | 1
  High Urea; >8.4 mmol/L | 56
  High Creatinine; ≥ 2.0 mg/dL | 8
  High Uric acid; >5.7 mg/dL | 9
  High Total Billirubin; > 1 mg/dL | 0
  High Creatinine Kinase; ≥ 170 U/L | 2
  High Serum Glucose Fasting; >118 mg/dL | 36
  High Serum Glucose Non-fasting; >118 mg/dL | 17
  High Cholesterol Total; > 220mg/dL | 131
  High Serum Calcium; >10.2 mg/dL | 5
  Low Serum Calcium; <8.6 mg/dL | 26
  High Serum Chloride; >108 mEq/L | 24
  Low Serum Chloride; <96 mEq/L | 36
  High Serum Potassium; >5.1 mEq/L | 36
  Low Serum Potassium; <3.3mEq/L | 11
  High Serum Sodium; > 145 mEq/L | 13
  Low Serum Sodium; < 133 mEq/L | 12
  Low Hematocrit; <37% | 21
  Low Hemoglobin; < 12 g/dL | 19
  High Leukocyte count; > 10.8 x 10^3 c/uL | 7
  Low Leukocyte count: < 4.8 x 10^3 c/uL | 4
  High Eosinophil count; > 5% | 3
  High Platelet count; >450 x 10^9 c/L | 0
  Low Platelet count; < 150 x 10^9 c/L | 1
  High Urine Protein; ≥ 2-unit increase | 2
  High Urine Glucose; ≥ 2-unit increase | 3

42. Secondary Outcome: Participants Who Died, Experienced Serious Adverse Events (SAEs), Adverse Events (AEs) or Discontinuations Due to AE During Treatment Beyond 140 Weeks
Description: as for outcome 28
Time Frame: Week 140 to Week 328
Population: Participants in France who completed the 130-week open-label extension phase and continued beyond Week 140 were included in safety sample.
Measure: Number; unit: Participants
Groups:
- Aripiprazole: Treatment beyond 140 weeks: Dosed at 2-15 mg/day (flexible dosing).
Arm/Group | Aripiprazole
Number analyzed (Participants) | 9
Participants
  Any AE | 7
  SAE | 1
  Death | 1
  Discontinuation due to AE | 3

ADVERSE EVENTS:
Arm/Group | 1 Double Blind Aripiprazole | 2 Double Blind Placebo | 3 Ext - Aripiprazole
Serious Adverse Events (participants affected / at risk) | 16/105 | 8/102 | 84/161
Other Adverse Events (participants affected / at risk) | 31/105 | 27/102 | 101/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Double Blind Aripiprazole (N=105) | 2 Double Blind Placebo (N=102) | 3 Ext - Aripiprazole (N=161)
ACQUIRED DIAPHRAGMATIC EVENTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 0 | 0 | 1
DEATH (General disorders) | 2 | 0 | 4
DIABETIC COMA (Nervous system disorders) | 0 | 0 | 1
ECZEMA VESICULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 3
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
FALL (Injury, poisoning and procedural complications) | 1 | 1 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 2
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0 | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 0 | 1
FAECALOMA (Gastrointestinal disorders) | 0 | 0 | 1
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
PSYCHOSOCIAL SUPPORT (Surgical and medical procedures) | 2 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
ASTHENIA (General disorders) | 0 | 0 | 2
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 10
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 0 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 3
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 1
MALAISE (General disorders) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 3
PYREXIA (General disorders) | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
EMBOLISM (Vascular disorders) | 0 | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 1
LETHARGY (Nervous system disorders) | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 4
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
SEPTIC SHOCK (Infections and infestations) | 1 | 0 | 0
VASCULAR DEMENTIA (Nervous system disorders) | 0 | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 2
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 0 | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 3
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 6
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1 | 0
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 1
SOCIAL PROBLEM (Social circumstances) | 0 | 0 | 1
SUDDEN CARDIAC DEATH (General disorders) | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 2
AGGRESSION (Psychiatric disorders) | 2 | 0 | 0
CATARACT (Eye disorders) | 1 | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 0 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
VARICOSE VEIN (Vascular disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 2
BRADYCARDIA (Cardiac disorders) | 1 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 3
CHEST PAIN (General disorders) | 0 | 1 | 0
CHILLS (General disorders) | 0 | 0 | 1
DEMENTIA (Nervous system disorders) | 0 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 0 | 3
MENDELSON'S SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 1
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
SUDDEN DEATH (General disorders) | 0 | 0 | 2
THROMBOSIS (Vascular disorders) | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Double Blind Aripiprazole (N=105) | 2 Double Blind Placebo (N=102) | 3 Ext - Aripiprazole (N=161)
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 10
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 10
SOMNOLENCE (Nervous system disorders) | 8 | 2 | 30
URINARY TRACT INFECTION (Infections and infestations) | 8 | 14 | 27
FALL (Injury, poisoning and procedural complications) | 3 | 4 | 18
INSOMNIA (Psychiatric disorders) | 2 | 4 | 14
ANXIETY (Psychiatric disorders) | 1 | 2 | 10
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 11
APATHY (Psychiatric disorders) | 0 | 0 | 13
DIARRHOEA (Gastrointestinal disorders) | 3 | 1 | 16
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 2 | 1 | 14
VOMITING (Gastrointestinal disorders) | 1 | 2 | 10
BRONCHITIS (Infections and infestations) | 4 | 3 | 27

LIMITATIONS AND CAVEATS:
Limitations of the study, such as early termination leading to small numbers of subjects analyzed and technical problems with measurement leading to unreliable or uninterpretable data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication